CLINICAL TRIAL: NCT02998138
Title: A Multi-center Study of Genomic and Psychological Factors Affecting Postoperative and Chronic Pain in Children Undergoing Invasive (Spine) Surgery
Brief Title: Postoperative and Chronic Pain Genetic Spine Surgery Study
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-8339; 2015-8633 (Other: CCHMC IRB)
Record Dates: First submitted 2016-03-07; First posted 2016-12-20 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Scoliosis; Kyphosis; Kyphoscoliosis
Keywords: Chronic Pain; Pain, Postoperative
MeSH Terms: conditions — Scoliosis; Kyphosis; Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be analyzed for a defined set of SNPs using PCR (TaqMan, ABI)/and Omni5M GWAS chip testing. DNA will be isolated from blood samples and also be used for pyrosequencing studies to obtain DNA methylation information for a specified set of genes or use of the MethylationEPIC array. The SNP sets were chosen using the adult studies cited in the Background and Significance section as evidence of potential importance. Given that the pain response in children and adolescents may involve a novel or different set of SNPs and additional SNPs of the above genes, the DNA samples gathered will be held for future analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
This will be an open label, prospective study to determine the association between specific genotypes, epigenetics and behavioral factors, with the phenotypes, defined by pain perception, postoperative pain, analgesic and side effect responses to perioperative opioids, chronic postoperative pain and gene expression in adolescents following major spine surgery.

DETAILED DESCRIPTION:
Safe and effective analgesia is an important unmet medical need in children. Despite efforts to promote non-pharmacologic interventions, drug treatment remains the standard of care for children experiencing severe pain following surgery. Inadequate pain relief after invasive surgery, and side effects from analgesics such as morphine occur frequently in up to 50% of children. A study of patient controlled analgesia (PCA) morphine use after spine surgery in adolescents observed a 45% incidence of postoperative nausea and vomiting and 7% incidence of respiratory depression. Presently, evidence-based dosing guidelines for opioid therapy have not been ascertained in the pediatric patient population, and remains a trial and error method. Despite aggressive pain management after spine surgery, findings showed that neither children's pain nor their analgesic use diminished significantly over time. As such, there is a critical knowledge gap in the medical literature that significantly impacts the pediatric pain management. Moreover, chronic postsurgical pain (CPSP, defined as pain attributable to the surgical procedure lasting for more than 2 months after surgery critically impacts 13-30% of children having surgery, and leads to chronic pain as adults imposing extraordinary annual costs on the health care system ($560-635 billion). It has been recently shown that pain unpleasantness predicts the transition from acute to moderate/severe persistent post-surgical pain, whereas anxiety sensitivity predicts the maintenance of moderate/severe post-surgical pain from 6 to 12 months after surgery. Spine fusion in adolescents is a particularly painful surgery with 15% incidence of pain even 5 years after surgery, and hence will serve as a good surgical model to evaluate the behavioral and genetic predictors of chronic postoperative pain. In recognition of this therapeutic challenge the investigators plan to evaluate the determinants of inter-individual differences in opioid analgesic responsiveness, adverse effects, pain perception and predictors of chronic postoperative pain in children.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 10 to 18, inclusive, years of age
2. Diagnosis of Idiopathic scoliosis, kyphosis and/or kyphoscoliosis
3. Scheduled for spine fusion.

Exclusion Criteria:

1. Patients on chronic pain medication (opioid use over 6 months prior to surgery)
2. Pregnant or breastfeeding females.
3. Children with a history of or active renal or liver disease.
4. Non-English speaking patients.
5. Developmental delay
6. Body Mass Index ≥ 30
7. Currently taking tricyclic, selective serotonin reuptake inhibitor (SSRI), serotonin-norepinephrine reuptake inhibitor (SNRI) class of medications (within the last month)
8. Cardiac conditions including, but not limited to, cyanotic heart disease, Hypoplastic Left Ventricle, arrhythmia, hypertension with ongoing treatment, Kawasaki Disease, cardiomyopathies. Patients with asymptomatic valvular lesions or defects may be included.
9. Severe lung disease such as cystic fibrosis, pulmonary fibrosis, pneumonia within the last month
10. History of seizures currently treated on medication (patients off medication and seizure free for greater than one year may be included)
11. Other known genetic diseases including but not limited to Ehlers Danlos, Downs' etc.
12. History of Obstructive sleep apnea by history (pauses during sleep, significant snoring, use of CPAP)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The investigators will recruit a total of 200 subjects over the study period to acquire the data necessary to derive a predictive model matching phenotype to genotype. They will be recruited from the population of children ages 10 to 18, inclusive, years scheduled for spinal surgical procedures.
Sampling Method: Non-Probability Sample
Enrollment: 880 (Estimated)
Dates: Start 2016-12; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) pain scores | Data will be collected for 48 hours postoperatively
Occurrences of respiratory depression | Data will be collected for 48 hours postoperatively
  Respiratory rate (RR) <10 on POD 1 and 2
Occurrences of post-operative nausea/vomiting (PONV) | Data will be collected for 48 hours postoperatively

SECONDARY OUTCOMES:
Amount of morphine (or equivalent) used by patient | Data will be collected for 48 hours postoperative
Chronic pain postoperatively | 2 - 6 months postoperatively
  Participants will complete questionnaires regarding pain since surgery was completed
Persistent pain postoperatively | 10 - 12 months postoperatively
  Participants will complete questionnaires regarding pain since surgery was completed
Opioid addiction by history on follow-up | 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Chidambaran, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (5):
- United States (5):
  - Stanford University Hospital, Stanford, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Duke Children's Hospital, Durham, North Carolina
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Narayanasamy S, Yang F, Ding L, Geisler K, Glynn S, Ganesh A, Sathyamoorthy M, Garcia V, Sturm P, Chidambaran V. Pediatric Pain Screening Tool: A Simple 9-Item Questionnaire Predicts Functional and Chronic Postsurgical Pain Outcomes After Major Musculoskeletal Surgeries. J Pain. 2022 Jan;23(1):98-111. doi: 10.1016/j.jpain.2021.06.014. Epub 2021 Jul 17. PMID 34280572